CLINICAL TRIAL: NCT04390204
Title: Evaluation of the Effect of a Postural Reflex Rehabilitation Program on a Foam Surface on Stress Urinary Incontinence in Women
Acronym: Protofoam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017/389/HP
Record Dates: First submitted 2020-05-06; First posted 2020-05-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Urinary Incontinence,Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Motor control exercises are performed on foam mats. The physiotherapist instructs them, and gives a description on paper, as well as a USB key allowing to view the exercises on video. A supervised home self-rehabilitation program on foam mats is implemented.
  Interventions: Other: intervenions
- control (No Intervention): According to the recommendations of learned societies, patients are offered voluntary MPP contraction work, in strength and endurance, in increasing complexity, under manual endocavitary control and under biofeedback. A supervised program of self-rehabilitation at home by voluntary contraction of MPP is set up.

INTERVENTIONS:
Other: intervenions — * Motor control exercises
  * A supervised home self-rehabilitation program
  Arms: Experimental

SUMMARY:
Urinary incontinence is defined by the International Continence Society as "any involuntary loss of urine complained by the patient". UI is a debilating condition affecting 25% to 45% of the female population. It is a recognized factor impairing the women's quality of life in women. Age, type and severity of UI as well as stress, fears and beliefs are variables that significantly affect the quality of life scores . Its costs are estimated at 2% of the health budget in European countries. Stress urinary incontinence (SUI) is characterized by a loss of urine that occurs with increased intra-abdominal pressure, such as coughing, laughing, sneezing, jumping, running, lifting loads or any other physical activity

. SUI accounts for 50% of UI types. For HAS (Haute Autorité de Santé), the first-line treatment is a conservative, non-medicinal and non-surgical treatment. Hay Smith's 2010 literature review concludes that pelvic floor muscle rehabilitation (PMP) must be the first-line treatment for SUI. However, there is a lack of evidence to define the best treatment regimen for PFM rehabilitation.

For 25 years, we have been performing assessment and rehabilitation programs for urinary incontinence. We see daily, as literature suggests, a link between continence and postural control. Previous studies, such as that we carried out within our service, tend to confirm the positive impact of reflex postural control on continence. Our team has already shown the feasibility of such a program and its effectiveness on stress urinary incontinence. Foam surfaces are devices used in the rehabilitation of reflex postural control. Several studies have shown that rehabilitation programs on foam surfaces improve reflex postural control better than the same exercises on stable ground. Smith et al. have shown impaired motor control of MPP on foam surfaces in women with stress urinary incontinence. However, the effect of a rehabilitation program with foam surface on urinary symptoms has never been evaluated.

For our main outcome, we propose to follow the recommendations of L. Rimstad in his recent prospective study of SUI assessment in 147 subjects aged 36 to 63 years, wich seems more in accordance with postural control disorder than the "gold standard" supine cough test wich has been found to have low sensitivity. The test pad on a trampoline allows to object a SUI in 91% of the negative patients to the test pad on firm surface. It therefore makes it possible to object stress urinary incontinence without invasive urodynamic investigations. It therefore seems justified for the comfort of our patients and the relevance of our results. The preliminary assessments and the skills of the physiotherapist make it possible to assess the patient's ability to perform this test. Our experience of carrying out trampoline tests or exercises for 25 years, as of the Rimstad team in the context of the treatment of SUI for 10 years, allows us to carry out this test in good conditions of efficiency , comfort and safety. Thus, we hypothesize that a rehabilitation program by supervised reflex postural control exercises on a foam surface can reduce the volume of urinary leakage in women. This study will also show the influence of such a program on symptoms and quality of life in women with urinary incontinence.

Innovative nature of our study We do not find in the literature any evaluation of the effectiveness of exercises on foam surface on stress urinary incontinence Our protocol, by its minimally invasive nature, would promote a better emotional experience for our patients Most studies in the context of incontinence are based on a semi-objective outcome assessment with symptoms questionnaire. We suggest using the short stress pad test, a more objective test for women, recommended by several authors We will observe the impact of our protocol on pelvic and low back pain, quality of life and any restrictions on social participations We hope to confirm the best acceptance of non-invasive treatments, without intravaginal probe in continence rehabilitation

Our protocol goes in the direction of:

* Literature reviews on urinary incontinence through supervised group sessions
* WHO's recommendations on the maintenance of balance and physical functions, and also the prevention of falls in adults

ELIGIBILITY:
Inclusion Criteria:

* 9≥18
* Patient with urinary incontinence according to the ICS criteria
* Patient affiliated to social security
* Patient having read and understood the information letter and signed the consent form
* Woman of childbearing age with effective contraception or menopausal status

Exclusion Criteria:

* Neurological, psychiatric and digestive pathology wich induces stress urinary incontinence
* Pregnant or parturient or lactating woman
* Person deprived of liberty by administrative or judicial decision or a person placed under the safeguard of justice, or guardianship or curatorship
* Anti-cholinergic treatment initiated less than 3 months ago
* Patient unable to complete the 15 planned visits to physiotherapist
* Patient participating in another clinical trial
* Patient unable to perform the first stress test pad
* No urinary leakage noted during the stress pad test (difference of weight before and after protection pad test = 0 g)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 88 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface to reduce stress urinary incontinence in women | through study completion, an average of 26 months
  difference in volume of urinary leaks before and after the supervised exercise protocol, measured during a standardized stress pad test

SECONDARY OUTCOMES:
Demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface on urinary symptoms | through study completion, an average of 26 months
  Urinary Symptom Profil (USP) questionnaire, higher scores mean a worse outcome (0-40).
Demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface on quality of life | through study completion, an average of 26 months
  The MOS 36-item short-form health survey (SF-36 questionnaire) + International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form ) ICIQ-SF (Scoring scale: 0-21) higher scores mean a worse outcome .
Demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface on improvement of urinary symptoms | through study completion, an average of 26 months
  Evaluation of the improvement of urinary symptoms using the Patient Global Impression of Improvement scale (PGI I) , higher scores mean a worse outcome (1-7).
Demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface low back pain | through study completion, an average of 26 months
  Assessment of low back pelvic pain using the Oswestry Disability Index questionnaire, higher scores mean a worse outcome (0-50).
emonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface on pelvic comfort | through study completion, an average of 26 months
  Evaluation of compliance with exercises and acceptance of treatment using the "compliance and acceptance" questionnaire
Demonstrate the effectiveness of a reflex postural control rehabilitation program with supervised exercises on a foam surface in terms of exercise compliance and acceptance of treatment | through study completion, an average of 26 months
  Pelvic comfort assessment using the Pelvic Floor Distress Inventory (PFID-20) questionnaire higher scores mean a worse outcome (0-80)

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Cabinet Rééducation Grabels, Grabels
  - cabinet de rééducation LINGOLSHEIM, Lingolsheim
  - Cabinet Rééducation Poitiers, Poitiers
  - CHU de ROUEN, Rouen
  - cabinet SCM feeling, Saint-Étienne-du-Rouvray

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322